CLINICAL TRIAL: NCT00762164
Title: Comparative Efficacy of a Vytorin 10/80 Tablet Split Into 4 (Estimated Dose Ezetimibe 2.5 + Simvastatin 20) Versus Simvastatin 20 Milligrams on LDL Cholesterol
Brief Title: Comparison of the Effect of Vytorin 10/80 Tablet Split Into 4 and Simvastatin 20 Milligrams on Low-density Lipoprotein (LDL) Cholesterol
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Bronx VA Medical Center (U.S. Federal Agency)
Responsible Party: Principal Investigator, Lawrence Baruch, Staff Physician, Bronx VA Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: VA---19-07-01
Record Dates: First submitted 2008-09-29; First posted 2008-09-30 (Estimated); Results first posted 2013-07-03 (Estimated); Last update posted 2013-07-03 (Estimated); Status verified 2013-04

CONDITIONS: Hypercholesterolemia
Keywords: Hypercholesterolemia; Statins; Ezetimibe
MeSH Terms: conditions — Hypercholesterolemia | interventions — Ezetimibe, Simvastatin Drug Combination; Simvastatin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1Vytorin 10/80 divided into 4 (Active Comparator): Vytorin 10/80 divided into 4
  Interventions: Drug: Vytorin
- Simvastatin (Active Comparator): Simvastatin 20 milligrams
  Interventions: Drug: Simvastatin

INTERVENTIONS:
Drug: Vytorin — Vytorin 10/80 split into 4
  Arms: 1Vytorin 10/80 divided into 4
Drug: Simvastatin — Simvastatin 20 milligrams
  Arms: Simvastatin

SUMMARY:
The purpose of this study is to compare the efficacy of a Vytorin 10/80 tablet, an approved agent for the treatment of elevated LDL cholesterol which combines the cholesterol absorption inhibitor Ezetimibe 10 mg and simvastatin 80 mg, when split into 4 using a tablet splitter, versus a whole simvastatin 20 milligram tablet.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with an LDL-cholesterol greater than 100 mg/dL
* Patients willing and able to provide signed informed consent

Exclusion Criteria:

* Patients receiving a statin (Lipitor, Crestor, Lescol, Simvastatin, or Pravachol)
* Patients intolerant of statins
* Patients receiving ezetimibe
* Patients intolerant of ezetimibe
* Patients receiving a niacin preparation
* Stroke, TIA, myocardial infarction, unstable angina, percutaneous coronary intervention, coronary artery bypass surgery, or major surgery within 3 months
* Cancer undergoing active treatment
* Creatinine clearance < 50 ml/minute
* Active liver disease or persistent elevation of SGOT or SGPT > 2 times the upper limit of normal level
* Participation in any clinical study within the last 30 days
* Drug addition or alcohol abuse within the past 6 months
* Use of azole antifungal agents, amiodarone, fibrates or immunosuppressant drugs within the last 3 months
* Active use of macrolide antibiotics or verapamil
* Consumption of grapefruit juice on a daily basis
* Patients unwilling or unable to provide informed consent
* Patients with poor compliance
* Women of childbearing potential

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2007-03; Primary Completion 2009-04 (Actual); Study Completion 2009-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lawrence Baruch, MD, Principal Investigator — Bronx VA Medical Center
Locations (1):
- Bronx VA Medical Center, The Bronx, New York, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Thirty-four patients were randomized from August 2007 through October 2008. Patients were recruited from our cardiology and lipid clinics.
Pre-assignment Details: There was no washout phase during the study. No patients were excluded after enrollment.
Period: Overall Study
Arm/Group | 1Vytorin 10/80 Divided Into 4 | Simvastatin
Started | 17 | 17
Completed | 14 | 15
Not Completed | 3 | 2
Not completed — Lost to Follow-up | 1 | 1
Not completed — Discontinued medication | 2 | 0
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 1Vytorin 10/80 Divided Into 4 | Simvastatin | Total
Number analyzed (Participants) | 17 | 17 | 34
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 13 | 11 | 24
  >=65 years | 4 | 6 | 10
Age Continuous [Mean (Standard Deviation); unit: years] | 55.3 (12.6) | 62.7 (7.8) | 59.1 (10.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 17 | 17 | 34
Region of Enrollment [Number; unit: participants]
  United States | 17 | 17 | 34

OUTCOME MEASURES:

1. Primary Outcome: LDL Cholesterol
Time Frame: 6 weeks
Measure: Mean (Standard Deviation); unit: % change in LDL cholesterol
Arm/Group | 1Vytorin 10/80 Divided Into 4 | Simvastatin
Number analyzed (Participants) | 14 | 15
% change in LDL cholesterol | -44.7 (19.0) | -27.1 (22.4)

2. Secondary Outcome: Total Cholesterol
Time Frame: 6 weeks
Measure: Mean (Standard Deviation); unit: % change in total cholesterol
Arm/Group | 1Vytorin 10/80 Divided Into 4 | Simvastatin
Number analyzed (Participants) | 14 | 15
% change in total cholesterol | -34.2 (13.0) | -19.9 (14.6)

ADVERSE EVENTS:
Time Frame: 6 weeks
Description: One patient never received the simvastatin in the simvastatin arm.
Arm/Group | 1Vytorin 10/80 Divided Into 4 | Simvastatin
Serious Adverse Events (participants affected / at risk) | 0/17 | 0/16
Other Adverse Events (participants affected / at risk) | 2/17 | 0/16
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 1Vytorin 10/80 Divided Into 4 (N=17) | Simvastatin (N=16)
Muscle pain-Myalgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No